CLINICAL TRIAL: NCT04614311
Title: Strategies Towards Personalised Treatment in Juvenile Idiopathic Arthritis (JIA): the MyJIA Trial.
Brief Title: Strategies Towards Personalised Treatment in Juvenile Idiopathic Arthritis (JIA).
Acronym: MyJIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Pernille Helen Bøyesen, MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 171224
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — triamcinolone hexacetonide

STUDY DESIGN:
Intervention Model Description: Parallel intervention were participants are assigned to either the control group or intervention group.
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates joints clinically will be blinded to study information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Intra-articular corticosteroid injections into active joints
  Interventions: Drug: Triamcinolone Hexacetonide 20 MG/ML
- Comparator (No Intervention): No intra-articular injections

INTERVENTIONS:
Drug: Triamcinolone Hexacetonide 20 MG/ML — JIA patients (age 1-18 years) starting TNFi treatment randomised to intervention will receive treatment with intra articular glucocorticoids (triamcinolone hexacetonide) injections in inflamed joints
  Other Names: Lederspan
  Arms: Intervention

SUMMARY:
Inhibitors of tumour necrosis factor (TNFa) reduce inflammation in patients with juvenile idiopathic arthritis (JIA), but only 20-40 percent achieve a state of no or very little disease activity. Tailored glucocorticoid joint injections are widely used (usually in general anaesthesia), but no controlled studies have addressed the effect of this approach. In Norway there are unique possibilities for early interventions, rapid escalation of medication and individualised therapy. The investigators aim to find the optimal ways to increase disease control and improve quality of life for JIA patients.

The hypothesis is that JIA patients starting TNF-inhibitors with added steroid injection of inflamed joints, will lead to improved outcomes compared to TNF-inhibitors with no joint injections, and that therapeutic drug monitoring, modern imaging and biologic and clinical profiling can be utilised to characterise JIA patients with different anti-TNF responses.

MyJIA is a national investigator initiated 48 weeks RCT of JIA patients starting TNF-inhibitors; 202 JIA patients will be randomised at baseline to A) concomitant intra-articular glucocorticoid injections versus B) no injections. Primary endpoint is the rate of sustained remission from weeks 24 to 36. Possible risk factors for not reaching remission will be analysed including clinical characteristics, drug antibodies/serum concentrations, patients' reported health status and preferences, molecular signalling (based on transcriptional, cellular and genetic risk) and synovitis detected by modern imaging (ultrasound and whole-body MRI).

Patients will be recruited from all Norwegian health regions through an established collaboration. Unit of Paediatric Rheumatology, Oslo University Hospital, with an extensive research track in this field, will be the coordinating centre. Broad research cooperation across disciplines is established. The trial is highly innovative in evaluating treatment options and strategies to individualise and optimise the efficacy and safety of JIA treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 1-18 years of age at the time of signing the informed consent.
2. Fulfilment of the International League of Associations for Rheumatology (ILAR) classification criteria for non-systemic JIA.
3. Clinical indication for starting TNFi treatment according to consensus between at least two physicians.
4. Naïve to TNFi or prior use of one TNFi (stopped at least 3 months before study inclusion and no previous TNFi treatment failure).
5. Juvenile Disease Activity Score (JADAS) >1 at baseline and at least one joint with active arthritis were joint injection is considered.
6. Willing to give written consent (participant ≥ 16, guardians if < 16 years of age, both participants and guardians if 16-18) and comply with the requirements of the study protocol.

Exclusion Criteria:

Medical Conditions

1. Major comorbidity including uncontrolled infectious, neurological or mental disease, malignant disease, severe heart failure, severe renal failure, active ulcus ventriculi, and uncontrolled diabetes mellitus.

   Prior/Concomitant Therapy
2. Used two or more TNFi.
3. Corticosteroid use (including i.a. injection) less than 4 weeks prior to randomisation.

   Other Exclusions
4. Known hypersensitivity to Triamcinolone hexacetonide (Lederspan) or any of the excipients (sorbitol, polysorbate or benzyl alcohol).
5. Concomitant therapy with CYP3A-inhibitors or digitalis glycosides.
6. Known inherited fructose intolerance
7. Presence of hepatitis B surface antigen (HBsAg) at screening.
8. Positive hepatitis C antibody test result at screening or within 12 months prior to starting study treatment.
9. Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (front), and TB testing. The choice of TB tests will be made by the investigator according to local licensing and standard of care.
10. Having received live vaccines less than two weeks prior to randomisation.
11. Drug / alcohol abuse which hampers adherence to the study protocol.
12. Language barriers that hampers adherence to the study protocol.
13. Pregnancy or breast-feeding.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 189 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
The proportion of JIA participants with sustained inactive disease | Week 24 to week 36.
  The proportion of participants with sustained, inactive disease from week 24 to week 36.
  Inactive disease is defined according the 2011 Wallace criteria:
  * No active arthritis†
  * Physician global assessment of disease activity score normal (0)
  * Erythrocyte sedimentation rate (ESR) within normal range
  * Morning stiffness ≤ 15 minutes
  * No active uveitis
  * No fever, rash, serositis, splenomegaly, or generalized lymphadenopathy attributable to JIA
  In addition, no use of any i.a. or p.o. corticosteroids from week 20 to week 36.
  †Active arthritis according to the ACR definition:
  1. a joint with swelling not due to bony enlargement OR, if no swelling is present
  2. limitation of motion accompanied by either pain on motion and/or tenderness.

SECONDARY OUTCOMES:
The proportion of participants with ACR pedi 30% response | Baseline to week 6,12 and 24
  American College of Rheumatology (ACR) paediatric 30% response (30% improvement in a minimum of 3 of any 6 variables in the paediatric core set criteria with no more than one of the remaining variables worsening more than 30%).
  Pediatric core set criteria:
  * Physician's global assessment of disease activity (visual analogue scale (VAS), range 0-100 where 0 represents best possible outcome).
  * Patient's/parent's global assessment of overall well-being (VAS, range from 0-100 where 0 represents best possible outcome)
  * Functional ability (Childhood Health Assessment Questionnaire, CHAQ, lower scores are indicative of better functioning)
  * Number of joints with active arthritis (range 0-71 where 0 represents best possible outcome)
  * Number of joints with limited range of movement (range 0-70 where 0 represents best possible outcome)
  * Erythrocyte sedimentation rate (normalised to a 0-10 scale where 0 represents best possible outcome)
The proportion of participants with ACR pedi 50,70 and 90% response | Baseline to week 6, 12 and 24.
  American College of Rheumatology (ACR) paediatric 50, 70 and 90% response (50,70 and 90% improvement in a minimum of 3 of any 6 variables in the pediatric core set (see above) criteria.
Juvenile arthritis disease activity score (JADAS) | Baseline to week 6, 12 and 24.
  The JADAS is a composite measure of disease activity with a range from 0 to 101 where 0 represents the best possible outcome and 101 the worst possible outcome.
  The JADAS is calculated as a sum of scores from:
  * Physician's global assessment of disease activity (visual analogue scale ranging from 0-100 where 0 represents best possible outcome and and 100 the worst possible outcome).
  * Patient's/parent's global assessment of overall well-being (visual analogue scale ranging from 0-100 where 0 represents best possible outcome and and 100 the worst possible outcome)
    - Erythrocyte sedimentation rate (ESR) (normalized to a 0-10 scale, according to the following formula: (ESR (mm/hour)-20)/10. 0 represents best possible outcome and and 10 the worst possible outcome)
  * Number of joints with active arthritis (range from 0 to 71 where 0 represents best possible outcome and and 71 the worst possible outcome)
Time to inactive disease | Baseline to 48 weeks
  Time (months) until participants reach inactive disease according to the Wallace criteria and JADAS.
Proportion of Participants with Minimal Disease Activity | Week 26 to 48
  Proportion of Participants with Minimal Disease Activity
Change from baseline in arthritis-related pain severity as measured by pain VAS item | 48 weeks
  Change from Baseline in Arthritis-Related Pain Severity as Measured by Pain Visual Analog Scale (VAS).
  The Pain VAS ranges from 0 to 100 where 0 represents no pain and 100 the worst possible level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pernille H Bøyesen, MD PhD, Study Director — Oslo University Hospital; Anna-Birgitte Aga, MD PhD, Principal Investigator — Oslo University Hospital; Berit Flatø, Prof, Principal Investigator — Oslo University Hospital
Locations (5):
- Norway (5):
  - Oslo University Hospital, Oslo, Oslo County
  - St Olavs Hospital, Trondheim, Trønderlag
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: No